CLINICAL TRIAL: NCT05563129
Title: The Importance of Teaching First Aid and Trauma Management to Primary School Students
Brief Title: Teaching First Aid and Trauma Management to School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Georgios Alexiou, Assistant professor, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 970/29-06-2021
Record Dates: First submitted 2022-09-24; First posted 2022-10-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Trauma-related Wound; Head Injury; Choking; Nose Bleed; Child, Only; Emergencies
Keywords: first aid training, children
MeSH Terms: conditions — Craniocerebral Trauma; Airway Obstruction; Epistaxis; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No first aid training (No Intervention)
- First aid training (Experimental)
  Interventions: Other: First aid lessons

INTERVENTIONS:
Other: First aid lessons — The school children will have first aid training
  Arms: First aid training

SUMMARY:
This proposal aims to describe research that will utilize first aid in primary education students and will attempt to identify the frequency with which the training should be repeated and the type of trainer who will carry out the training program.

DETAILED DESCRIPTION:
The training concerns courses with theoretical knowledge and practical skills related to first aid. Taking into account children's cognitive and psychological development, students will be trained in the following topics: calling an ambulance, managing bleeding, handling an unconscious patient, drowning, and managing a head injury. Classroom teachers and specialized staff will teach classes. The evaluation of knowledge and skills will be done with a questionnaire. The evaluation will take place before and immediately after the training, two months and seven months after the training.

ELIGIBILITY:
Inclusion Criteria:

* Students at primary schools and kindergarten, 4-9 years old

Exclusion Criteria:

* Students over 9 years old

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Number of participants that know first aid | 1 day pre the training
  We will use questionnaire to assess this outcome
Number of participants that learnt first aid | 1-day post the training
  We will use questionnaire to assess this outcome
Comparing the results of the training about the facilitators' performance | 2 months post the training
  We will use questionnaire to assess this outcome
Number of participants that retain the first aid knowledge | 7 months post the training
  We will use questionnaire to assess this outcome

CONTACTS AND LOCATIONS:
Locations (1):
- George Alexiou, Ioannina, Greece